CLINICAL TRIAL: NCT04696029
Title: Phase II Trial of Eflornithine/DFMO as Maintenance Therapy for Molecular High Risk/Very High Risk and Relapsed/Refractory Medulloblastoma
Brief Title: DFMO as Maintenance Therapy for Molecular High/Very High Risk and Relapsed Medulloblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC016
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Difluoromethylornithine (DFMO) (Experimental): study subjects will receive 730 Days of oral difluoromethylornithine (DFMO) at a dose of 2500 mg/m2 BID on each day of study.
  Interventions: Drug: Difluoromethylornithine

INTERVENTIONS:
Drug: Difluoromethylornithine — DFMO (difluoromethylornithine is an inhibitor of ornithine decarboxylase (ODC) designated chemically as 2-(difluoromethyl)-DL-ornithine monohydrochloride monohydrate.
  The dosage form to be used in this study is provided as a convex tablet containing 192 mg eflornithine (equivalent to 250 mg of eflornithine HCl, monohydrate). The tablets are packaged and sealed in opaque white HDPE bottles, and each bottle contains 100 tablets. The DMFO tablets are supplied by USWorldMeds (USWM).
  The tablets are to be stored at room temperature (20-250C).
  Other Names: Eflornithine; DFMO

SUMMARY:
Difluoromethylornithine (DFMO) will be used in an open label, multicenter, study as Maintenance Therapy for Molecular High Risk/Very High Risk and Relapsed/Refractory Medulloblastoma.

DETAILED DESCRIPTION:
In this study subjects will receive 730 Days of oral difluoromethylornithine (DFMO) at a dose of 2500 mg/m2 BID on each day of study.

Subjects will be evaluated in 3 Cohorts:

Cohort 1: Molecular High Risk Medulloblastoma Cohort 2: Molecular Very High Risk Medulloblastoma Cohort 3: Relapsed/Refractory Medulloblastoma

A total of 118 subjects across all cohorts will be enrolled to ensure that there will be 107 evaluable subjects (32-39 per cohort)

ELIGIBILITY:
Inclusion Criteria:

1. Age: 0-21 years of age at diagnosis
2. Pathology All patients must either have a pathologically confirmed diagnosis of medulloblastoma with molecular grouping identified by either Nanostring or methylation profiling.

   Cohort 1- Molecular High Risk:
   * Metastatic non-MYC amplified Group 3
   * Metastatic Group 4
   * Metastatic non-WNT/non-SHH (Must be non-MYC amplified)

   Cohort 2- Molecular Very High Risk
   * Metastatic OR MYCN amplified OR TP53 mutant non-infant (>3 yrs) SHH
   * MYC amplified Group 3
   * Non-WNT, non-SHH infant (< 3 yrs)

   Cohort 3: Relapsed/Refractory Medulloblastoma
3. Pre-enrollment tumor survey:

   Prior to enrollment on this study, a determination of mandatory disease staging must be performed:
   * Tumor imaging studies including: Brain and spine MRI
   * Lumbar Puncture only if previously positive
   * Bone Marrow aspiration/biopsy only if previously positive
   * This disease assessment is required for eligibility and preferably should be done within 2 weeks prior to first dose of study drug, but must be done within a maximum of 4 weeks before first dose of study drug.
4. Disease Status: Subjects must have no evidence of disease, or stable* residual nonbulky** disease.

   *Stable residual disease defined as non-progression over 2 separate imaging studies at least 6 weeks apart

   **Non-bulky disease defined as maximal cross-sectional area < 3cm^2 at enrollment. Patients with leptomeningeal disease are allowed to participate on study.
5. Timing from prior therapy:

   Enrollment (first dose of DFMO) no later than 60 days after last dose of conventional chemotherapy. Patients who have undergone high dose chemotherapy (HDCT) with autologous stem cell transplantation (SCT) are eligible if more than 45 days have elapsed since date of last SCT.
6. Patients must have a Lansky or Karnofsky Performance Scale score of ≥ 50% (see Appendix II) and patients must have a life expectancy of ≥ 2 months.
7. All clinical and laboratory studies for organ functions to determine eligibility must be performed within 7 days prior to first dose of study drug unless otherwise indicated below.
8. Patients must have adequate organ functions at the time of registration:

   * Hematological: Hematological recovery as defined by ANC ≥750/μL, platelets ≥30 (non-transfused x 7 days)
   * Liver: Adequate liver function as defined by AST and ALT <10x upper limit of normal
   * Renal: Adequate renal function defined as (perform one of the following): Creatinine clearance or radioisotope GFR ≥ 70 mL/min/1.73 m2 or a serum creatinine based on age/gender
9. Females of childbearing potential must have a negative pregnancy test. Patients of childbearing potential must agree to use an effective birth control method. Female patients who are lactating must agree to stop breast-feeding.
10. Written informed consent in accordance with institutional and FDA guidelines must be obtained from all subjects (or patients' legal representative).

Exclusion Criteria:

1. BSA of <0.25 m2
2. Metastatic disease outside of CNS
3. Relapsed/refractory patients who are radiation-naïve and age 5 years or older at time of enrollment
4. Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.
5. Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the hematological and bone marrow suppression effects of prior chemotherapy.
6. Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
7. Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with event free survival (EFS) during study | 2 years plus 5 years follow up
  o To evaluate the efficacy of difluoromethylornithine (DFMO) as a single agent in preventing relapse in patients with molecular high risk and very high risk medulloblastoma, and relapsed/refractory medulloblastoma based upon the 2-year progression-free survival rate (PFS) compared to relevant historical controls.

SECONDARY OUTCOMES:
Length of time that participants experience Overall Survival (OS) | 7 years
  o To evaluate the efficacy of difluoromethylornithine (DFMO) as a single agent in patients with molecular high risk and very high risk medulloblastoma, and relapsed/refractory medulloblastoma based upon overall survival
Determine the Overall Response Rate (ORR) of Participants using Modified RANO Criteria | 2 years
  To evaluate the efficacy of difluoromethylornithine (DFMO) as a single agent in patients with molecular high risk and very high risk medulloblastoma, and relapsed/refractory medulloblastoma based upon Response Rate for patients with non-bulky residual disease present.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years plus 30 days
  To develop a complete safety and tolerability profile of difluoromethylornithine (DFMO) in pediatric and young adult subjects with medulloblastoma.
Determine amount of DFMO in the CSF at 3 hours post dose | 2 years
  o To measure CSF penetration after DFMO administration in pediatric subjects with medulloblastoma

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Huang, MD, Study Chair — Beat Childhood Cancer
Locations (23):
- United States (22):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Rady Children's Hospital, San Diego, California
  - Stanford University, Stanford, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - All Children's Hospital Johns Hopkins Medicine, St. Petersburg, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Advocate Aurora Research Institute, Chicago, Illinois
  - Kentucky Children's Hospital, Lexington, Kentucky
  - Norton Children's Research Institute/Affiliated with University of Louisville School of Medicine, Louisville, Kentucky
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Levine Children's Hospital, Charlotte, North Carolina
  - Randall Children's Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Children's Blood and Cancer Center, Austin, Texas
- CHUQ, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beat Childhood Cancer Consortium website — https://research.beatcc.org/